CLINICAL TRIAL: NCT01628835
Title: Low Glycemic Index Diet Intervention on Insulin Resistance of Overweight Pregnant Women.
Brief Title: Low Glycemic Index (GI) Diet Management for Pregnant Woman With Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Kunshan City Maternal and Child Health (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Weili Yan, Professor, Director, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: version1.0; NSFC 81273168 (Other Grant/Funding Number: National Science Fundation of China)
Record Dates: First submitted 2012-05-10; First posted 2012-06-27 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Overweight; Pregnant Women
Keywords: overweight; pregnancy; diet counselling; glycemic
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dietary glycemic index diet (Experimental): Based on the national diet and physical activity recommendations for pregnant women (total energy intake, protein and vitamin etc.), counseling for a low dietary glycemic index diet will be provided.
  Interventions: Behavioral: Low dietary glycemic index diet
- National recommendation diet (Active Comparator): Provision of food and dietary counseling according to the national prenatal nutrition recommendation without GI information
  Interventions: Behavioral: National recommendation diet

INTERVENTIONS:
Behavioral: Low dietary glycemic index diet — Based on the national diet and physical activity recommendations for pregnant women (total energy intake, protein and vitamin etc.), counseling for a low dietary glycemic index diet will be provided
  Arms: Low dietary glycemic index diet
Behavioral: National recommendation diet — Provision of food and dietary counseling according to the national prenatal nutrition recommendation without GI information
  Other Names: recommended diet for pregnant women
  Arms: National recommendation diet

SUMMARY:
The study is a randomized, single-blinded, controlled intervention trial to compare the effect of a low glycemic index diet versus diet recommended by the Chinese Dietary Guide for Pregnant Women on maternal and neonatal insulin resistance and adverse gestational events.

DETAILED DESCRIPTION:
Overweight in pregnant women increases maternal insulin resistance and risk of adverse pregnancy outcomes. Recent evidence from both animal studies and human subject studies shows that adverse environmental exposures during pregnancy result in adverse influence on offsprings. The hypothesis of the current study is that the healthy intervention during pregnancy to overweight pregnant women--low glycemic diet, may improve the maternal and neonatal insulin resistance at birth.

The current study adopts randomized, single-blinded, controlled intervention trial, gives low glycemic index diet intervention based on the national diet and physical activity recommendations for pregnant women to the intervention group and only national diet recommendations to the control group. Four diet consultation interviews will be done,at baseline (first prenatal examination), the end of the 1st trimester, the 2nd trimester and the 3rd trimester respectively, including diet assessment and diet consultation specifically to adopting low glycemic diet. Glycemic load of diet will be calculated based on 24 hour diet recall data for each individual at every visit to help to lower their diet glycemic load by modifying some daily foods. The effect of intervention is investigated by comparing the insulin resistance levels between the two arms at birth and when infants are at age 2. For discrete traits, such as incidence of gestational diabetes and gestational hypertension, Person's chi-square tests were used. For continuous traits, such as insulin resistance index, maternal weight gain and neonatal birth weight, we use t-tests for comparisons between two groups. The study expects that long-term low GI diet intervention have beneficial effects on controlling maternal and neonatal insulin resistance to overweight women and long term health.

ELIGIBILITY:
Inclusion

* Singleton pregnancy;
* Pregnant women with BMI≥24 kg/m2 at first antenatal examination;
* aged 18 years to 45 years;
* The week of first prenatal examination equal to or less than 12 weeks;
* Take routine prenatal examination;
* Willing and able to give informed consent. Exclusion
* Artificial impregnation;
* History of hypertension, diabetes, coronary heart disease or mental disorder;
* With Special diet habit(e.g. vegetarianism/ veganism).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2012-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maternal insulin resistance | During pregnancy
Cord blood C-peptide | at delivery
Maternal weight gain | measured before delivery
  measured before delivery (minus pre-conceptual body weight)
Incidence of gestational diabetes | during pregnancy
  from 1st antenatal visit to delivery
Incidence of macrosomia | at delivery
  birth weight >= 4000g

SECONDARY OUTCOMES:
Incidence of gestational hypertension | during pregnancy
  proportion of patients with SBP/SBP>=140/90 for 3 visits
Mean infant birth weight | at delivery
cesarean | at delivery
head circumference | at delivery
Mean gestational age | at delivery
Incidence of premature delivery | at delivery
  gestational age <37 week at delivery

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Kunshan Maternal and Child Health Care Hospital, Kunshan, Jiangsu
  - International Peace Maternity and Child Care Centers of Communications University, Shanghai

REFERENCES:
- [Derived] Zhang Y, Wang L, Yang W, Niu D, Li C, Wang L, Gu P, Xia Y, Shen Y, Yan J, Zhao Q, Mu K, Yan W. Effectiveness of Low Glycemic Index Diet Consultations Through a Diet Glycemic Assessment App Tool on Maternal and Neonatal Insulin Resistance: A Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Apr 18;7(4):e12081. doi: 10.2196/12081. PMID 30998227